CLINICAL TRIAL: NCT00859846
Title: Comparison of Ultrasound Guided Arterial Line Placement in Long Axis Versus Short Axis in Pediatric Patients.
Brief Title: Ultrasound Guided Arterial Line Placement in Long Axis Versus Short Axis in Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2340
Record Dates: First submitted 2009-03-09; First posted 2009-03-11 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: General Anesthesia
Keywords: Arterial line; Ultrasound; Anesthesia; Pediatric

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Long Axis arterial line placement (Experimental): Twenty four patients will undergo arterial line placements using long axis arterial line placement under ultrasound.
  Interventions: Procedure: Arterial line placement
- Short Axis arterial line placement (Experimental): Twenty four patients will undergo arterial line placements using short axis arterial line placement under ultrasound.
  Interventions: Procedure: Arterial line placement
- Palpation arterial line placement (Active Comparator): Twenty four patients will undergo arterial line placements using Traditional palpation arterial line placement.
  Interventions: Procedure: Arterial line placement

INTERVENTIONS:
Procedure: Arterial line placement — The following measures will be collected and compared.
  1. Time (in seconds) required for successful placement of the arterial line. This is the time elapsed between either palpation or placement of ultrasound probe on the patient's wrist and the successful demonstration of arterial waveform on the anesthesia monitor.
  2. number of attempts, defined as forward advancements of needle, required to cannulate the artery.
  3. number of separate skin punctures.
  4. number of arteries into which entry is attempted.
  Other Names: Ultrasound guided (short vs Long axis)

SUMMARY:
The use of ultrasound is becoming widespread to guide the placement of arterial lines for both vascular access and regional anesthesia in the field of anesthesia. Arterial line placement can be challenging, especially in the pediatric population. Frequently multiple attempts are required with relatively high failure rates. This can result in excessive needle punctures and extended OR times. A few studies have looked at the use of ultrasound to decrease OR time and increase success rates both in adult and pediatric populations. These studies compared the traditional palpation method with either short axis or long axis views of the vessel using ultrasound guidance. No study to date has compared short axis and long axis views for arterial line placement in either the pediatric or adult population. Our study compares success rates and OR times when long and short axis methods of arterial line insertion are employed in the pediatric population.

DETAILED DESCRIPTION:
An Arterial line is an intraoperative monitor that is frequently placed in the pediatric population. Due to their smaller anatomy and more compliant skin, arterial lines can be more difficult to insert in the pediatric population than in adults. Additionally, lower perfusion pressure and larger subcutaneous adipose tissue can make pulse palpation more difficult. Ultrasound is a modality that can directly image the radial, ulnar, or brachial artery. Along with 2D ultrasound, doppler ultrasound can be utilized to confirm that an artery is not a vein. Once the vessel is identified, the vessel can be viewed in either the long or short access. The ultrasound beam is only 1 millimeter thick so a practitioner must stabilize the probe to view the vessel, especially in the long axis view. Once the artery is viewed in long axis, the needle can be directly visualized all the way into the vessel. Visualization of a guidewire or catheter in the vessel can confirm proper arterial access. In a short access ultrasound view, it is possible to see tissue movement and sometimes a hyperechoic (bright) dot which represents the needle. Tissue movement can help confirm the needle is immediately above the artery at all times. The advantage of the short axis view is that less precision is needed to hold and position the transducer than with the long axis view. The disadvantage of the short axis view is that the operator cannot see the tip of the angiocatheter as it enters the vessel. As a result, the proximal portion of the angiocatheter can be above the artery but the distal tip could be to the side of the artery.

ELIGIBILITY:
Inclusion Criteria:

* The investigators will identify patients 0 to 14 years of age who are classified as ASA physical status ≤4 and scheduled to have surgery under general anesthesia

Exclusion Criteria:

* History of vasculitis, autoimmune disease, Reynauds phenomenon or disease
* History of no collateral perfusion
* The absence of an upper extremity artery to cannulate such as a bilateral amputee
* A child in DHS custody
* Infection at the site of insertion
* Patient refusal.

Ages: 1 Day to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 29 (Actual)
Dates: Start 2009-03-17 (Actual); Primary Completion 2018-09-25 (Actual); Study Completion 2018-09-25 (Actual)

PRIMARY OUTCOMES:
Using the long axis ultrasound view increases the success rate of arterial line insertions compared to using the short axis view. | 1.5 year
  Using the long axis ultrasound view increases the success rate of arterial line

SECONDARY OUTCOMES:
Using the short axis view, when successful, results in quicker insertion than when using the long axis view. | 1.5 year
  Using the short axis view, when successful, results in quicker insertion than when using the long axis view.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto J de Armendi, MD, Principal Investigator — Oklahoma University Health Sciences Center
Locations (1):
- The University of Oklahoma Health Sciences Center Deparment of Anesthesiology, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schwemmer U, Brederlau J. [Ultrasound techniques in anesthesiology--guided vascular access using sonography]. Anasthesiol Intensivmed Notfallmed Schmerzther. 2006 Nov;41(11):740-9. doi: 10.1055/s-2006-958847. German. PMID 17151988
- [Background] Shiver S, Blaivas M, Lyon M. A prospective comparison of ultrasound-guided and blindly placed radial arterial catheters. Acad Emerg Med. 2006 Dec;13(12):1275-9. doi: 10.1197/j.aem.2006.07.015. Epub 2006 Nov 1. PMID 17079789